CLINICAL TRIAL: NCT04449822
Title: Emergency Surgery Versus Colorectal Stents for the Management of Malignant Colonic Obstructions: a Prospective Cohort Study
Brief Title: Emergency Surgery Versus Colorectal Stents for the Management of Malignant Colonic Obstructions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zaza Demetrashvili (Other)
Responsible Party: Sponsor-Investigator, Zaza Demetrashvili, Associate Professor, Surgery Department, Tbilisi State Medical University
Organization: Tbilisi State Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07122017
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer
Keywords: Hartmann's procedure, colostomy, colonic stenting.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency surgery (Active Comparator): Surgical decompression with colostomy with or without resection and eventual re-anastomosis.
  Interventions: Procedure: Emergency surgery
- Colonic stenting (Active Comparator): The colonic stent placement
  Interventions: Procedure: Colonic stenting

INTERVENTIONS:
Procedure: Emergency surgery — Surgical decompression with colostomy with or without resection and eventual re-anastomosis.
  Arms: Emergency surgery
Procedure: Colonic stenting — The colonic stent placement to relieve the colonic obstruction.
  Arms: Colonic stenting

SUMMARY:
The study evaluates and compares effect of emergency surgery and colonic stents for treatment of malignant colonic obstructions.

DETAILED DESCRIPTION:
Acute colonic obstruction is one of the common clinical presentations of colorectal cancer. Surgical decompression with colostomy with or without resection and eventual re-anastomosis is the treatment of choice; however, emergency surgery is associated with higher morbidity and mortality.

The colonic stent insertion effectively decompressed the obstructed colon and avoid needs of emergency surgery. This method is a palliation and bridge to surgery. Colonic stents allowed surgery to be performed electively.

ELIGIBILITY:
Inclusion Criteria:

* Patient with malignant colorectal obstructions.
* Patient's approval to participate in the study.

Exclusion Criteria:

* Patient's preference for either treatment method.
* Patient's refusal to participate in the study.
* Patients in the ASA group 4 and 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
The time of clinical relieve of obstruction | 24 hours after surgery/procedure

SECONDARY OUTCOMES:
Stent related complications | time of hospital stay, an average 10 day.
  perforation, migration, stent obstruction
Mortality | 30 day after surgery/procedure
  30-day mortality
Blood loss | time of surgery/procedure
  Blood loss during emergency surgery or during colonic stenting.
operation time | during surgery/procedure
  duration of surgery/procedure
Overall complications | 30 day after surgery/procedure
  complications which developed in postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Zaza Demetrashvili, Principal Investigator — Tbilisi State Medical University
Locations (1):
- Tbilisi State Medical University, Tbilisi, Yes, Georgia

REFERENCES:
- [Result] Merabishvili G, Agdgomelashvili I, Mosidze B, Demetrashvili Z. Emergency surgery versus colorectal stenting for the management of left-sided malignant colon obstructions:A prospective cohort study. Acta Scientific Medical Sciences 2021, 5(4):18-23. doi: 10.31080/ASMS.2020.05.0863